CLINICAL TRIAL: NCT01122745
Title: Comparison of Pain Relief After Single Shot Interscalene Block With Continuous Interscalene Block for Arthroscopic Rotator Cuff Shoulder Surgery: A Randomized Study
Brief Title: Single Shot vs Continuous Interscalene Block for Rotator Cuff Repair
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-243-B
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Pain; Rotator Cuff; Surgery
Keywords: continuous block; single shot; interscalene; rotator cuff surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Catheter Group: Patient will have continuous interscalene block for pain relief placed preoperatively. They will go home with the portable pump. Pain score will be tracked via phone and compared with the control or single short group.
- Single shot group: Patient will have single shot interscalene block and will go home. Pain will be tracked using phone. Pain will be compared with the catheter group.

SUMMARY:
1. Rotator cuff have painful post surgery recovery.
2. Single shot interscalene with oral analgesics may or may not be enough
3. Continuous nerve block may be too much for the surgery
4. The idea is to compare two techniques to see if the two techniques can improve patient pain control and satisfaction.

DETAILED DESCRIPTION:
After consent patients will be randomized to one of the two groups: Control Group or the Experimental Group. Patients will be blinded to the group assignment.

In the Control Group the patient will be given single shot interscalene block using ultrasound technique following established guidelines. The procedure will be done after starting intravenous access and placing standard anesthesia monitors (EKG, Blood Pressure Cuff and Pulse-Ox) on the patient. Following accepted aseptic guidelines the nerves will be visualized at the base of the neck using ultrasound machine. Once proper nerve roots or trunks visualized 3 mg/kg of 0.5 % bupivacaine will be injected in small blouses.

In the Experimental Group, after placement of monitors, the nerves will be visualized using ultrasound machine. There after a catheter will be placed. They subjects will be dosed using 0.5% bupivacaine 3 mg/kg for the surgery via the catheter.

The extent of block before the surgery will be evaluated at 30 minutes post injection. Surgery will be done with sedation. Conversion of anesthetic technique to general anesthesia will be considered failure of the technique to provide adequate surgical anesthesia.

At the end of the case the patient will be taken to recovery and will be evaluated for pain. If patient is having pain of 3 or more then they will be treated as follows.

In single shot group will be offered to be blocked again or treated with oral narcotics.

In the catheter group patient will be dosed with 10 ml 1% lidocaine. If it fails to provide any relief then the catheter will be pulled back and another 10 ml1% lidocaine will be given. If still not effective then it will be replaced. Refusal of patient to replace the catheter will result in patient dropping out of the study.

Working catheter will be left in place for at least 48 hrs. Patients will be allowed to take oral pain medicines as prescribed by their surgeons. The patient will be sent home with pain pump to continuously give them 0.125% bupivacaine at 5 ml per hr with an option to get extra dose of 5 ml q hr if needed. The pain control will be monitored by phone daily till catheter comes out.

ELIGIBILITY:
Inclusion Criteria:

* adult
* rotator cuff surgery
* agreeing to regional block for pain control

Exclusion Criteria:

* pregnancy
* neuropathy
* any allergies to local anesthetics
* any contraindication to nerve blocks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All pateint undergoing arthroscopic rotator cuff surgrey and agreed to have regional block for pain control
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2010-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
pain relief | 2-3 days
  Patients having rotator cuff repair surgery will be randomized to either single shot or continuous catheter group. Pain score will be followed for 2 days to see which group gets better pain relief.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Hospitals, Chicago, Illinois, United States